CLINICAL TRIAL: NCT03831828
Title: Retrospective Study of Gene Status and Clinical Outcome of Esophageal Squamous Cell Carcinoma(ESCC).
Brief Title: Correlation of Gene Status and Clinical Outcomes in ESCC
Acronym: ESCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: LiuJunFeng (Other)
Collaborators: OrigiMed (Industry)
Responsible Party: Sponsor-Investigator, LiuJunFeng, Director of thoracic surgery, Hebei Medical University Fourth Hospital
Organization: Hebei Medical University Fourth Hospital (Other)
Other Study IDs: HebeiMUFH-ESCC
Record Dates: First submitted 2019-02-04; First posted 2019-02-06 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2018-09

CONDITIONS: Prognosis of Patients With ESCC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Lymph node metastasis Positive: good prognosis; without Lymph node metastasis.
- Lymph node metastasis Negative: poor prognosis; with Lymph node metastasis.

SUMMARY:
The incidence of esophageal squamous cell carcinoma is highly regional and familial. The current treatment plan is based on the stage and location of the tumor.By studying the relationship between the status of different genes and prognosis, it can help doctors to develop precise and individualized treatment plans.

ELIGIBILITY:
Inclusion Criteria:

* Esophageal cancer patients who underwent surgery treatment, and postoperative pathological diagnosis was squamous cell carcinoma. Patients with ESCC have complete clinical information.

Exclusion Criteria:

* Patients who also suffering from other tumors.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Taihang Mountain area population in northern China.
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2018-12-26 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Gene test | 2019-2 to 2019-4
  466 Tumor-associated gene test by next-generation sequencing(NGS)

CONTACTS AND LOCATIONS:
Locations (1):
- Junfeng Liu, Shijiazhuang, Hebei, China